CLINICAL TRIAL: NCT06885021
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Trial to Evaluate the Safety and Efficacy of HDM1002 Tablets in Chinese Overweight and Obese Adults
Brief Title: Evaluate the Safety and Efficacy of HDM1002 Tablets in Chinese Overweight and Obese Adults
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HDM1002-301
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HDM1002 tablets 200mg once daily (Experimental): HDM1002 200mg, oral, once daily, 52weeks
  Interventions: Drug: HDM1002 200mg, oral, once daily, 52 weeks
- HDM1002 tablets 400mg once daily (Experimental): HDM1002 400mg, oral, once daily, 52weeks
  Interventions: Drug: HDM1002 400mg, oral, once daily, 52 weeks
- Placebo (Placebo Comparator): HDM1002 placebo, oral, once daily, 52weeks
  Interventions: Drug: HDM1002 placebo, oral, once daily, 52 weeks

INTERVENTIONS:
Drug: HDM1002 200mg, oral, once daily, 52 weeks — HDM1002 200mg, oral, once daily, 52 weeks
  Arms: HDM1002 tablets 200mg once daily
Drug: HDM1002 400mg, oral, once daily, 52 weeks — HDM1002 400mg, oral, once daily, 52 weeks
  Arms: HDM1002 tablets 400mg once daily
Drug: HDM1002 placebo, oral, once daily, 52 weeks — HDM1002 placebo, oral, once daily, 52 weeks
  Arms: Placebo

SUMMARY:
A Phase 3 Trial to Evaluate the Safety and Efficacy of HDM1002 Tablets in Overweight and Obese Adults

ELIGIBILITY:
Inclusion Criteria:

* BMI≥28 but < 40.0 kg/m2 at screening or randomization，or BMI≥24.0 kg/m2 but < 28 kg/m2 with any of the following:

  1. Hypertension
  2. Dyslipidemia
  3. Obstructive sleep apnea syndrome
  4. MASH
  5. Pain in the weight-bearing joints
* At least one previous failure to lose weight through lifestyle modification was defined as < 5% weight loss after ≥3 months of lifestyle modification

Exclusion Criteria:

* Weight change ≥5% as reported or documented.
* Previous diagnosis of type 1, type 2, or any other type of diabetes.
* Diagnosis of overweight or obesity due to other diseases or medications.
* History or family history of medullary thyroid carcinoma, C cell hyperplasia, or multiple endocrine neoplasia type 2.
* Have diseases or conditions that affect gastric emptying or gastrointestinal absorption of nutrients, such as bariatric surgery or other gastrectomy, irritable bowel syndrome, dyspepsia, chronic pancreatitis, etc. Or a history of acute pancreatitis or acute gallbladder disease within 3 months before signing ICF.
* GLP-1R agonist use within 6 months prior to signing ICF.
* Use of hypoglycemic drugs within 3 months before signing ICF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Estimated)
Dates: Start 2025-03-28 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage Change From Baseline in Body Weight | 44weeks
  Weight was recorded in kilograms (kg), and accuracy to the nearest 0.1 kg,
Percentage Change of Participants Achieving Weight Loss ≥ 5% | 44weeks
  Weight was recorded in kilograms (kg), and accuracy to the nearest 0.1 kg

SECONDARY OUTCOMES:
Percentage Change of Participants Achieving Weight Loss ≥ 10% and ≥ 15% | 44weeks
  Weight was recorded in kilograms (kg), and accuracy to the nearest 0.1 kg.
Change From Baseline in Waist Circumference | 44 weeks, 52 weeks
  Waist Circumference was recorded in cm
Percentage Change of Participants Achieving Weight Loss ≥ 5% , ≥ 10% and ≥ 15% | 52 weeks
  Weight was recorded in kilograms (kg), and accuracy to the nearest 0.1 kg.

IPD SHARING:
Plan to Share IPD: Undecided